CLINICAL TRIAL: NCT00555477
Title: Aromatase Inhibitors in Premenopausal Breast Cancer Patients With Chemotherapy-Induced Ovarian Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped after 69 subjects were enrolled because of poor accrual.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Lynn Henry, Principal Investigator, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.044; HUM 12443 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: premenopausal breast cancer with chemotherapy-induced ovarian failure
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anastrozole (Experimental)
  Interventions: Drug: anastrozole

INTERVENTIONS:
Drug: anastrozole — 1 mg tablet by mouth once a day
  Other Names: Arimidex

SUMMARY:
Women with hormone-receptor positive breast cancer are typically treated with hormone therapy as part of their treatment after surgery. In the past few years it has been found that treatment with aromatase inhibitors is superior to tamoxifen in postmenopausal women. Tamoxifen is still used for premenopausal women, however, because aromatase inhibitors are not effective in women who have functioning ovaries. Some women are premenopausal at the time they are diagnosed with breast cancer, but then stop having menstrual periods when they are treated with chemotherapy. It is unclear if these women can also be treated safely with aromatase inhibitors.

In this clinical trial the researchers will try to answer this question. Women with hormone receptor positive breast cancer who become postmenopausal with chemotherapy will be invited to participate in this study. Each woman will be treated with one of the aromatase inhibitors, anastrozole (Arimidex), and then carefully monitored to ensure that her ovaries do not start making estrogen. If her estrogen level remains low, then she will continued to be followed for 18 months. If the level increases to the level typically seen in premenopausal women, however, then she will stop taking part in this study.

The study will also evaluate multiple factors that may help doctors predict who will tolerate the therapy without having their ovaries start making estrogen again. Some of the factors to be evaluated include other hormone levels (blood tests) as well as family history of early menopause (mother, sisters). In addition, changes in certain genes that affect how patients' bodies handle chemotherapy drugs will be tested to see if they affect whether or not patients recover ovarian function. Overall, the purpose of the study is to determine which patients who become postmenopausal from chemotherapy are likely to tolerate aromatase inhibitor treatment safely, and how often the patients' ovarian function needs to be tested during treatment.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study:

1. You must be at least 18 years of age and not older than 60 years of age
2. You have breast cancer which was confined to the breast and lymph nodes under the arm, and have no evidence of cancer elsewhere
3. You must have had surgical removal of your tumor, and if indicated, radiation therapy must have been completed or planned
4. Your tumor must express estrogen and/or progesterone receptors
5. You must have had a menstrual period within 6 months before starting chemotherapy for your breast cancer.
6. You must have been treated with a chemotherapy regimen that includes cyclophosphamide (Cytoxan). Your menstrual periods must have stopped for at least 8 weeks starting during or after chemotherapy.

Exclusion Criteria:

You are not eligible to participate in this study if:

1. Your ovaries have been surgically removed, treated with radiation therapy, or if you are taking medications (Zoladex™ or Lupron™) to block the function of your ovaries.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L. Henry, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Result] Henry NL, Xia R, Banerjee M, Gersch C, McConnell D, Giacherio D, Schott AF, Pearlman M, Stearns V, Partridge AH, Hayes DF. Predictors of recovery of ovarian function during aromatase inhibitor therapy. Ann Oncol. 2013 Aug;24(8):2011-6. doi: 10.1093/annonc/mdt149. Epub 2013 Apr 23. PMID 23613476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the University of Michigan, the Dana-Farber Cancer Institute, and Johns Hopkins University from 2008 until 2010.
Pre-assignment Details: 69 patients were enrolled however only 59 patients began treatment with anastrozole. Patients that were enrolled and found to have estradiol concentrations greater than 20 pg/ml were not treated.
Groups:
- Anastrozole Part 1: In the initial version of the clinical trial (designated part 1), subjects were required to have serum estradiol and FSH (Follicle-stimulating hormone) concentrations within the postmenopausal range according to local institutional guidelines within 28 days of enrollment. Subjects taking tamoxifen at the time of screening were only required to have postmenopausal serum estradiol concentrations. Subjects were treated with anastrozole, 1 mg orally daily.
- Anastrozole Part 2: During the conduct of the trial the study was amended to change the eligibility criteria because of difficulties with the estradiol assay. Subjects enrolled after the amendment were required to sign consent and then have an average baseline estradiol concentration of ≤20 pg/ml in order to be considered eligible.
Period: Overall Study
Arm/Group | Anastrozole Part 1 | Anastrozole Part 2
Started | 14 | 45
Completed | 12 | 32
Not Completed | 2 | 13
Not completed — Adverse Event | 0 | 9
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: Initiated treatment with Anastrozole, 1 mg orally daily.
Groups:
- Anastrozole Part 1: In the initial version of the clinical trial (designated part 1), subjects were required to have serum estradiol and FSH concentrations within the postmenopausal range according to local institutional guidelines within 28 days of enrollment. Subjects taking tamoxifen at the time of screening were only required to have postmenopausal serum estradiol concentrations. Subjects were treated with anastrozole, 1 mg orally daily.
- Anastrozole Part 2: Analysis of the first 18 subjects enrolled revealed a greater than expected discontinuation of AI therapy because of elevated serum estradiol concentrations. Discontinuation was believed to be primarily due to greater than expected variability in the assay as opposed to true recovery of ovarian function. Therefore, the protocol was amended. Subjects with an average baseline estradiol concentration of ≤20 pg/ml were considered eligible for part 2 and initiated treatment with anastrozole 1 mg orally daily.
- Total: Total of all reporting groups
Arm/Group | Anastrozole Part 1 | Anastrozole Part 2 | Total
Number analyzed (Participants) | 14 | 45 | 59
Age, Continuous [Median (Full Range); unit: years] | 46 [44 to 52] | 50 [40 to 56] | 50 [40 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 45 | 59
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 45 | 59

OUTCOME MEASURES:

1. Primary Outcome: The Number of Women Who Recover Ovarian Function Within 12 Months of Al Monotherapy
Description: In part 1 ovarian function recurrence is defined as one estradiol value >20 pg/ml or two consecutive values >10 pg/ml. In part 2 ovarian function recurrence is defined as a >75% increase in estradiol levels over prior if prior value was 15-30 pg/ml, or one estradiol value >30 pg/ml, or three consecutive values >20 pg/ml.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Anastrozole Part 1 | Anastrozole Part 2
Number analyzed (Participants) | 14 | 45
participants | 8 | 13

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) will be captured while each patient is taking study medication and for 30 days after the patient discontinues study medication and/or trial participation.
Arm/Group | Anastrozole
Serious Adverse Events (participants affected / at risk) | 2/59
Other Adverse Events (participants affected / at risk) | 53/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=59)
Infection Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=59)
Fatigue (General disorders) | 14 (15)
Insomnia (Psychiatric disorders) | 15 (16)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 5 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (7)
Hot flashes/flushes (Vascular disorders) | 18 (19)
Hemorrhage, Vagina (Reproductive system and breast disorders) | 8 (10)
Edema: limb (General disorders) | 8 (8)
Joint-function (Musculoskeletal and connective tissue disorders) | 8 (8)
Musculoskeletal/Soft Tissue - Other (Specify) (Musculoskeletal and connective tissue disorders) | 6 (9)
Dizziness (Nervous system disorders) | 5 (7)
Mood alteration (Nervous system disorders) | 4 (4)
Mood alteration (Nervous system disorders) | 11 (12)
Neuropathy: sensory (Nervous system disorders) | 7 (8)
Pain-Abdomen (General disorders) | 6 (7)
Pain-Breast (Reproductive system and breast disorders) | 4 (5)
Pain-Limb (Musculoskeletal and connective tissue disorders) | 8 (9)
Pain-Head (Nervous system disorders) | 4 (4)
Pain-Joint (Musculoskeletal and connective tissue disorders) | 23 (29)
Pain-Muscle (Musculoskeletal and connective tissue disorders) | 7 (8)
Pain - Other (Specify) (General disorders) | 4 (6)
Vaginal dryness (Reproductive system and breast disorders) | 14 (15)

LIMITATIONS AND CAVEATS:
Because of poor accrual, the trial was closed after 69 of a planned 150 patients were enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No